CLINICAL TRIAL: NCT05312086
Title: Prospective Analysis of Quantitative and Qualitative Muscle Abnormalities in Children With X-linked Hypophosphatemia (XLH)
Brief Title: Muscle Abnormalities in Children With XLH
Acronym: MDmuscleXLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A01386-33
Record Dates: First submitted 2022-01-24; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-01

CONDITIONS: Muscle Weakness; XLH
Keywords: XLH rickets; IMAT; intraMAT; muscle weakness; MRI
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with X-linked hypophosphatemic (Other): Patient group composed of 10 patients aged between 5 to 17 years old, female or male, with X-linked hypophosphatemic (XLH) rickets, severity of clinical and radiological damage (pain, muscle weakness and severe bone deformities) and ongoing growth (lesser bone age than 15 years old), child under conventional treatment
  Interventions: Other: MRI
- healthy volunteers (Other): control group composed of 20 helthy volunteers aged between 5 to 17 years old, female or male, without any endocrine pathology, not suffering from XLH, matching by age (+/- 6 months) and sex
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Performing the muscle MRI requires the cooperation of the child in order to remain lying down and motionless throughout the duration of the MRI, about 45 minutes.
  Performing MRI does not require the injection of contrast products or radiopharmaceuticals.

SUMMARY:
XLH rickets is a rare disease with muscle weakness. Fat parameters such as IMAT and intraMAT could be increased in this disease. IMAT and intraMAT will be calculated on MRI for 11 XLH children versus 20 typically developing children. The investigator will compare the percentage of IMAT in the XLH group versus control group and the difference concerning the intraMAT between the two groups.

DETAILED DESCRIPTION:
Single-center, prospective, non-randomized, controlled study with XLH and healthy volunteer children.

This study involves performing muscle MRI in healthy child volunteers to assess and compare the structure and composition of muscles to those of muscles in children with XLH pathology (muscle MRI of XLH patients is performed as part of standard medical care).

During this study we will have two groups: XLH group and a control group with typically developing children. In the XLH group, composed of 10 patients aged between 5 ans 17 years, female or male and ongoing growth (lesser bone age than 15 years old), have XLH and the most severe radiological deformities,clinical complications (pain and muscular weakness), have already done a muscle MRI of the lower limb during their follow-up.

The control group composed of 20 healthy volunteers aged between 5 ans 17 years old, female or male and without any endocrine pathology. A muscle MRI is necessary for healthy volunteers.

Every child will be alone After signing the informed consent by the 2 parents, the patient or the healthy volunteer and his parents, the MRI assessment will be performed on the same day.

Performing the muscle MRI requires the cooperation of the child in order to remain lying down and motionless throughout the duration of the MRI, i.e. approximately 45 minutes.

Performing MRI does not require the injection of contrast products or radiopharmaceuticals.

ELIGIBILITY:
Inclusion Criteria common criteria to the 2 groups:

* Age: between 5 and 17 years.
* Sex: male or female.
* Informed consent, signed by both parents or holder of parental autority after being informated of the study.
* Affiliation to a social security schema or having the right to.

Inclusion criteria for XLH Patients :

* Patient suffer of X-linked hypophosphatemia rickets.
* Severity of clinical and radiological damage (pain, muscle weakness and severe bone deformities).
* Growth in progress (bone age less than 15 years).
* Child under conventional treatment: patient responding to conventional treatment or
* under treatment with Burosumab (patient in treatment failure under treatment conventional).

incluion criteria for helthy volunteers :

* Healthy voluntary subjects, not suffering from XLH.
* Matching by age (+/- 6 months) and sex.

Exclusion Criteria common to the 2 groups :

* Not being able to stay still during the MRI examination (approximately 45 min).
* Growth completed.
* History of lower limb surgery.
* Contraindications to MRI
* Holders of parental authority under AME.
* Holders of parental authority under tutorship / curatorship.

Exclusion criteria for Healthy volunteers :

* Patients with endocrine, contracted or muscular pathology.
* Patient receives a long-term treatment.
* Patients with a high athletic level.
* BMI-IOTF <20 or> 27.8

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Quantify and compare muscle composition in XLH children versus healthy control children to demonstrate a link between muscle function and muscle quality. | 1 day
  calculation of inter-muscular adipose tissue will be done in cm2

SECONDARY OUTCOMES:
Measurement of muscle strength on force platforms, during gait analysis. Power test by mechanography of the jump (bipod and monopodal). Grasping test and correlation of fatty infiltration and functional data. | 1 day
  The Outcome Measure is BMI (Kg/m²)
Quantitative analysis of the muscles of the lower limbs (volume and length) | 1 day
  The Outcome Measure is BMI (Kg/m²)